CLINICAL TRIAL: NCT01016431
Title: Effects of Atrial Rate-adaptive Pacing on Exercise Capacity in Patients With Chronic Heart Failure Complicated by Chronotropic Incompetence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Prof. Serafino Fazio, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHRON-INC-09
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-11

CONDITIONS: Heart Failure; Exercise Tolerance
Keywords: cardiac pacing; heart failure; oxygen consumption; ventricular dysfunction; left, exercise tolerance; chronotropic incompetence; pacemaker programming
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rate adaptive (Experimental): Patients will have their ICD programmed in a AAI-R mode, with peak atrial rate set at 85% of age-adjusted predicted maximal HR
  Interventions: Other: Rate-adaptive pacemaker programming
- Control (Active Comparator): ICDs will be programmed in the usual VVI backup pacing mode at 40 bpm
  Interventions: Other: VVI at 40 bpm

INTERVENTIONS:
Other: Rate-adaptive pacemaker programming — The ICD will be programmed in a AAI-R mode, with peak atrial stimulation rate set at 85% of maximal predicted heart rate, and ongoing protection VVI backup at 40 bpm
  Arms: Rate adaptive
Other: VVI at 40 bpm — ICDs will be programmed in VVI mode at 40 bpm
  Arms: Control

SUMMARY:
Chronotropic incompetence consists of an insufficient increase in heart rate during effort, and its presence is recognized as a common feature in patients with heart failure due to left ventricular systolic dysfunction, apparently suggesting a worse prognosis. Little is known about the possible benefits of its reversal in such patients.

The investigators working hypothesis is that the modulation of chronotropic response, as obtained by means of atrial rate-adaptive pacing may improve functional capacity in persons with chronic heart failure and chronotropic incompetence.

To explore this hypothesis,the investigators will enroll 20 patients with NYHA II/III heart failure, low left ventricular ejection fraction (<40%) and chronotropic incompetence (Maximal heart rate <80% of predicted value in a symptom-limited incremental test), who already underwent implantation of dual-chamber implantable defibrillator for prevention of sudden cardiac death. The study will have a randomized, double-blind, cross-over design.

The procedures, to be carried out at one month from each reprogramming (VVI backup pacing vs. AAI-R "active" pacing), will comprise: blood sampling for NT-proBNP, incremental symptom-limited cardiopulmonary exercise testing (CPX), constant-workload cardiopulmonary test (50% of max WR), quality-of-life questionnaire, 24-hour ECG monitoring.

The primary end-point will be peak oxygen consumption on CPX. Secondary end-points will include acute response to reprogramming, and data derived from constant-WR tests, Holter monitoring and QoL.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II/III chronic heart failure on optimal medical therapy
* Sinus Rhythm
* Left ventricular ejection fraction less than 40 %
* Chronotropic incompetence on maximal exercise testing (maximum heart rate < 80% of predicted value)
* Age 18-75
* carrier of dual chamber ICD device
* Informed Consent

Exclusion criteria:

* Unable to perform cardiopulmonary exercise testing (for any reason)
* Absolute contraindication to maximal exercise testing
* Moderate to severe anemia (Hb<10 g/dL)
* Diagnosis of Sick Sinus Syndrome or high-degree atrioventricular block
* recent hospitalization for acute decompensated heart failure (<1 month)
* recent acute coronary syndrome (<3 months)
* Active neoplastic disease
* Active myocarditis / endocarditis
* Acute decompensated heart failure during study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen consumption on cardiopulmonary exercise testing | 1 month

SECONDARY OUTCOMES:
Peak Heart Rate on Cardiopulmonary exercise testing | 1 month
Quality of life as assessed by Minnesota Living with Heart Failure and SF-36 Questionnaires | 1 month
Heart Rate Variability on Holter Monitoring | 1 month
Acute Change in Peak Oxygen Consumption after reprogrammation | 1 hour
NT-proBNP levels | 1 Month

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University - Department of Internal Medicine, Naples, Italy